CLINICAL TRIAL: NCT02998190
Title: A Randomised, Double-Blind, Placebo-Controlled Study of a Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) of a FimH Antagonist, EB8018, in Healthy Volunteers.
Brief Title: First-in-Human Single and Multiple Dose of EB8018
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enterome (Industry)
Collaborators: Quotient Clinical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EBFIM116
Record Dates: First submitted 2016-12-13; First posted 2016-12-20 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Single oral dose of EB8018 (Experimental): Single ascending doses, sequential group design
  Interventions: Drug: Single Ascending Doses of EB8018
- Single oral dose of placebo (Placebo Comparator): Single doses, matching placebo
  Interventions: Drug: Single Ascending Doses of placebo
- Multiple oral doses of EB8018 (Experimental): Multiple ascending doses, daily for 14 days
  Interventions: Drug: Multiple Ascending Doses of EB8018
- Multiple oral doses of placebo (Placebo Comparator): Multiple ascending doses, daily for 14 days
  Interventions: Drug: Multiple Ascending Doses of placebo

INTERVENTIONS:
Drug: Single Ascending Doses of EB8018
  Arms: Single oral dose of EB8018
Drug: Single Ascending Doses of placebo
  Arms: Single oral dose of placebo
Drug: Multiple Ascending Doses of EB8018
  Arms: Multiple oral doses of EB8018
Drug: Multiple Ascending Doses of placebo
  Arms: Multiple oral doses of placebo

SUMMARY:
The purpose of this study is to determine the safety profile of single and multiple doses of EB8018 in healthy male subjects, to determine the pharmacokinetic profile of single and multiple doses of EB8018 in healthy male subjects and to assess preliminary effects of EB8018 on the healthy male gut microbiome.

DETAILED DESCRIPTION:
Crohn's Disease is a chronic inflammatory disease of the gastrointestinal tract. Emerging evidence suggests that the microbiome plays an important role in triggering an abnormal mucosal immune response in patients with Crohn's Disease. Independent studies have demonstrated an imbalance of the microbiome with a significant increase of E coli with invasive properties, termed adherent-invasive E coli (AIEC). These AIEC bacteria attach to the gut wall of susceptible patients via the fimbrial adhesion protein FimH, and subsequently trigger inflammation by invading and proliferating within the gut wall. EB8018 is an oral small molecule that is designed to block FimH thereby preventing the entry of AIEC into the gut wall thereby disarming the bacteria without disrupting the gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Age ≥ 18 to ≤ 55 years of age
* Body mass index of 19.0 to 30.0 kg/m2
* Normal ECG, showing no clinically relevant deviations, as judged by the investigator (QTcF ≤450 ms)

Exclusion Criteria:

* Subjects who have received any Investigational Medicinal Product in a clinical research study within the previous 3 months.
* History of any drug or alcohol abuse in the past 2 years
* Regular alcohol consumption in males >21 units per week
* Current smokers and those who have smoked within the last 12 months
* Positive drugs of abuse test result
* Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever, even inactive, is not allowed.
* Chronic infection or acute significant infection or fever within the previous 5 weeks prior to the start of IMP administration
* Malignancy or prior malignancy, with a disease-free interval of less than 5 years after diagnosis and intervention

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Number of Treatment Related Adverse Event, including Abnormal Laboratory Events to evaluate the safety and tolerability profile of single ascending and multiple ascending doses of EB8018 compared with placebo in healthy subjects | Between screening and 7-10 days after the last dose
  The variables for analysis will be the difference of EB8018 compared with placebo for incidence, severity and type of adverse events, including changes in vital signs, physical examinations, laboratory safety tests and ECGs

SECONDARY OUTCOMES:
The amount of EB8018 in plasma | Between Day 1 predose and 48 hours after the (last) dose
  To characterize the amount of EB8018 in plasma over time - pharmacokinetics (PK) - after a single oral dose and multiple oral doses in healthy subjects
The amount of EB8018 in urine | Between Day 1 predose and 48 hours after the (last) dose
  To characterize the amount of EB8018 in urine over time - pharmacokinetics (PK) - after a single oral dose and multiple oral doses in healthy subjects
The amount of EB8018 in stool | Between predose and 48 hours after the (last) dose
  To characterize the amount of EB8018 in urine over time - pharmacokinetics (PK) - after a single oral dose and multiple oral doses in healthy subjects
Analysis of microbiome richness | Between predose and 48 hours after the (last) dose
  To compare the abundance of gene richness, all phyla and certain species such as E. Coli

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Clinical, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No